CLINICAL TRIAL: NCT05400954
Title: Association of Silicone Breast Implant Reconstruction and -Enlargement With Overall Wellbeing, Lymphoma and Auto-immune Disease - Breast Implant Illness
Brief Title: Association of Silicone Breast Implants With Overall Wellbeingand Auto-immune Diseases
Acronym: AREOLA-B
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Erasmus Medical Center (Other); Maastricht University Medical Center (Other); Zuyderland Medical Centre (Other); Medisch Spectrum Twente (Other); Ziekenhuisgroep Twente (Other); Velthuis Kliniek (Unknown)
Responsible Party: Principal Investigator, Sanne Schagen, Prof. Dr., The Netherlands Cancer Institute
Other Study IDs: M21REO
Record Dates: First submitted 2022-05-27; First posted 2022-06-02 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer; Breast Implant; Complications; Autoimmune Diseases
Keywords: Silicone Breast Implant; Breast Reconstruction; Breast Cancer; Breast Implant Illness; Autoimmune disease
MeSH Terms: conditions — Breast Neoplasms; Autoimmune Diseases | interventions — Mammaplasty; Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Reconstruction with silicone breast implant: The cohort will be composed of women who underwent surgery for first invasive breast cancer or ductal carcinoma in situ (DCIS) in the years 2000 to 2015 in the collaborating centres. Eligible for inclusion in the exposed group are all women who underwent (i) mastectomy followed by immediate implant-based reconstruction, (ii) mastectomy followed by implant-based reconstruction at a later stage and (iii) latissimus dorsi flap reconstruction with a silicone breast implant
  Interventions: Procedure: Breast reconstruction with silicone breast implant
- Breast cancer surgery without silicone breast implant: . Eligible for inclusion in the comparison group are women who underwent (i) simple mastectomy without reconstruction, (ii) autologous reconstruction and (iii) breast conserving surgery. From the latter group a frequency-matched sample will be selected based on age at breast cancer diagnosis and calendar year of diagnosis.
  Interventions: Procedure: Breast conserving surgery/Mastectomy/Autologous reconstruction
- cosmetic breast augmentation: . Women who underwent cosmetic augmentation in the years 2000 to 2015 constitute a second comparison group. From this group a frequency-matched sample will be selected based on age and year of surgery.
  Interventions: Procedure: Breast Augmentation

INTERVENTIONS:
Procedure: Breast reconstruction with silicone breast implant — (i) mastectomy followed by immediate implant-based reconstruction, (ii) mastectomy followed by implant-based reconstruction at a later stage and (iii) latissimus dorsi flap reconstruction with a silicone breast implant.
  Other Names: Breast Reconstruction
  Groups: Reconstruction with silicone breast implant
Procedure: Breast conserving surgery/Mastectomy/Autologous reconstruction — (iv) simple mastectomy without reconstruction, (v) autologous reconstruction and (vi) breast conserving surgery,
  Groups: Breast cancer surgery without silicone breast implant
Procedure: Breast Augmentation — (vii) cosmetic augmentation with silicone breast implants
  Groups: cosmetic breast augmentation

SUMMARY:
Background: Implant-based breast reconstructions contribute considerably to the quality of life of breast cancer patients. A knowledge gap exists concerning the potential role of breast implants in the development of so called 'breast implant illness' and autoimmune diseases in breast cancer survivors with a silicone breast implant-based reconstruction. Breast implant illness is a constellation of non-specific symptoms reported by a small group of women with silicone breast implants.

Methods/Design: The Areola study is a multi-centre historic cohort study with prospective follow-up aiming to assess the risk of 'breast implant illness' and autoimmune diseases in female breast cancer survivors with and without silicone breast implants. The cohort consists of breast cancer survivors who received surgical treatment with silicone implant-based reconstruction in six major hospitals across the Netherlands in the period between 2000 and 2015. As comparison group, a frequency-matched sample of breast cancer survivors without breast implants will be selected. An additional group of women who received breast augmentation surgery in the same years will be selected to compare their characteristics and health outcomes with those of breast cancer patients with implants. All women still alive will be invited to complete a web-based questionnaire covering various health related topics. The entire cohort including deceased women will be linked to the population based computerized databases of Statistics Netherlands. These databases include a registry of diagnostic codes, a pharmacotherapeutic prescriptions registry and a cause-of-death registry in which diagnoses of autoimmune diseases will be identified. Outcomes of interest are the prevalence and incidence of BII and the prevalence and incidence of autoimmune diseases. In addition, risk factors for the development of BII and autoimmune disorders will be assessed among women with implants.

Discussion: The Areola study will contribute to the availability of reliable information on the risks of breast implant illness and autoimmune diseases in Dutch breast cancer survivors with silicone breast implants. This will inform breast cancer survivors and aid future breast cancer patients and their treating physicians to make informed decisions about reconstructive strategies after mastectomy.

Keywords: Silicone breast implants, Breast reconstruction, Breast cancer, Breast Implant Illness, Autoimmune disease

DETAILED DESCRIPTION:
There are various indications for implantation of a silicone breast implant. Most frequently, silicone breast implants are used in breast augmentation procedures for cosmetic reasons. In the field of oncology, breast implants are used for reconstructive purposes after mastectomy in the context of breast cancer treatment or prevention. A small percentage of breast reconstructions are performed in women with a hereditary predisposition for breast cancer who undergo bilateral prophylactic mastectomy. In the Netherlands, every year approximately 20,000-30,000 silicone breast implants are inserted for cosmetic (70%) and reconstructive purposes (30%)

From the 1990s onwards, there has been discussion in the scientific community about possible health risks associated with silicone breast implants. It was hypothesised that silicone breast implants could be the cause of breast cancer and sarcoma due to induction of pre-neoplastic fibrotic scar tissue. Furthermore, a variety of auto-immune-, auto-inflammatory- and neurological disorders have been attributed to silicone breast implants. The debate has generated significant research into potential cancer risks from silicone breast implants. Already in the 1990s, results from this research led to rejection of the hypothesis about associations between silicone breast implants and carcinoma or sarcoma of the breast. Most of the other alleged associations between silicone breast implants and various diseases were also discarded due to a lack of evidence after multiple epidemiologic investigations with long-term follow-up. A number of high-powered studies did suggest evidence for an association between silicone breast implants and autoimmune diseases.. However, these studies suffered from a number of methodological shortcomings such as failure to control for confounders, relying solely on unconfirmed patient-reported data, uncertainty as to which participants had silicone implants and high loss to follow-up. These caveats made their conclusions ultimately unconvincing. A strong causal association with silicone breast implants has only been established for Anaplastic Large Cell Lymphoma of the breast, an extremely rare T-cell lymphoma that can develop in the implant capsule.

In contrast to expectations based on the current body of scientific evidence, a number of women reports various health issues following placement of a silicone breast implant. These complaints are generally nonspecific and not attributable to one organ system. Reported symptoms include among others: numbness and tingling of the extremities, joint pain, myalgia, hair loss, cognitive problems, sicca complaints, chronic fatigue, rashes and hives, food intolerances and excessive sweating. The interval between placement of silicone breast implants and the onset of symptoms varies greatly from patient to patient. 'Autoimmune Syndrome Induced by Adjuvants' (ASIA) and 'Silicone Implant Incompatibility Syndrome' are two of the different names that have been coined to describe this constellation of symptoms. Lately, use of the term 'Breast Implant Illness' (BII) has become more commonplace among patients and patient advocates22. In line with difficulty in defining the diagnosis of this entity, its aetiology is unclear. The idea has been postulated that in susceptible individuals, silicone micro-particles that are shed from the implant set into motion a complex mechanism of immune dysregulation via receptor and cytokine pathways. However, so far an exact biochemical mechanism has not been described. With regard to the treatment of BII, suggestive evidence exists that explantation of the implant leads to an improvement of symptoms in at least part of affected women. However, two small observational studies from the Netherlands and the United States did not observe a statistically significant difference in the prevalence of BII-associated symptoms between women with cosmetic silicone breast implants and appropriate comparison groups. These results cast doubts with regard to an association between silicone breast implants and complaints ascribed to BII. In the absence of proof of proportionate organic abnormalities in patients with BII complaints, explanations from a behavioural science perspective have also been put forward, considering the role that psychological and social mechanisms can play in amplification of functional somatic symptoms 28. Striking similarities exist between the typical symptoms ascribed to BII and disorders like chronic fatigue syndrome and fibromyalgia.

With increasing evidence demonstrating the positive impact of breast-contour preserving surgical strategies on quality of life, a growing group of breast cancer patients undergo implant-based breast reconstructions after mastectomy. International data show an upsurge in immediate breast reconstruction over the past decade with rates now reaching around 50% in both The United States and England. Most breast cancer patients undergoing mastectomy are candidates for reconstruction. Although patient preference increasingly plays a role in the choice for a specific reconstructive strategy, factors such as patient's BMI, smoking, comorbidities or available surgical expertise may limit the options. In the Netherlands, the vast majority (83,4%) of immediate breast reconstructions are implant-based with the proportion of autologous reconstructions being around 11% 37. International trends also indicate a shift towards implant based reconstructions.

The current position of the U.S. Food and Drug Administration is that silicone breast implants are safe and reliable devices when used as labelled. Although the purported association between silicone breast implants and autoimmune diseases has been investigated many times, this issue has not been definitively resolved. Large epidemiologic studies investigating the potential association between silicone breast implants and the controversial new entity referred to as BII are lacking. Elucidating the role of implants in autoimmune disease and BII is of great importance to breast cancer patients who often have to make decisions about undergoing an implant-based reconstruction in a short timeframe. Uncertainty fuelled by lay reports on unsubstantiated side effects of silicone breast implants can complicate the decision-making process for patients as well as healthcare professionals. Possibly, this may lead to patients opting for more technically and physically demanding alternatives such as autologous reconstructions which entail longer recovery times, a higher risk of complications and higher expenses 40.

The Areola study is a Dutch prospective cohort study aiming to assess the risk of BII and autoimmune diseases in female breast cancer survivors with and without silicone breast implants. Focussing on sound epidemiological method, it attempts to overcome limitations that hampered previous studies. An additional goal is to identify risk factors for the development of BII and autoimmune disorders among women with implants. The Areola study was set up to meet the demand for reliable information about the role of silicone breast implants on long-term health outcomes in breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* surgery for first invasive breast cancer or ductal carcinoma in situ (DCIS) in the years 2000 to 2015 in the collaborating centres

Exclusion Criteria:

* above the age of 60 at breast cancer diagnosis
* above the age of 80 years at time of inclusion
* Not residing in Netherlands

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women who underwent surgery for first invasive breast cancer or ductal carcinoma in situ (DCIS) in the years 2000 to 2015 in the collaborating centres. Eligible for inclusion in the exposed group are all women who underwent (i) mastectomy followed by immediate implant-based reconstruction, (ii) mastectomy followed by implant-based reconstruction at a later stage and (iii) latissimus dorsi flap reconstruction with a silicone breast implant. Eligible for inclusion in the comparison group are women who underwent (i) simple mastectomy without reconstruction, (ii) autologous reconstruction and (iii) breast conserving surgery. From the latter group a frequency-matched sample will be selected based on age at breast cancer diagnosis and calendar year of diagnosis. Women who underwent cosmetic augmentation in the years 2000 to 2015 constitute a second comparison group. From this group a frequency-matched sample will be selected based on age and year of surgery.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Breast Implant Illness | 20years
  Relative risk (RR) of experiencing the following complaints in exposed and comparison groups:
  Cognitive impairment joint pain myalgia anxiety feeling depressed skin rashes weakness sleeping problems headache hair loss food intolerances and allergies numbness/tingling in upper and lower limbs dry eyes morning stiffness night sweats heart palpitations shoulder pain
Autoimmune disease | 20years
  Relative risk (RR) and Incidence rate (IR) for the following illnesses in exposed group and comparison group:
  Sjögren's Syndrome (SjS) Rheumatoid Arthritis (RA) Systemic Lupus Erythematosus (SLE) Systemic Sclerosis (SSc), Mixed Connective Tissue Disease (MCTD) Antiphospholipid Syndrome (APS) Ankylosing Spondylitis Sarcoidosis Multiple Sclerosis (MS) hypothyroidism hyperthyroidism psoriatic disease inflammatory bowel disease fibromyalgia chronic fatigue syndrome irritable bowel syndrome
Relative risk to develop autoimmune diseases and BII complaints associated with certain risk factors: | 20years
  RR for BII and autoimmune diseases will be assessed associated with riskfactors in the domains of demographics, lifestyle, reproductive history, medical- and treatment history and family history. Furthermore the influence of psychosocial factors like satisfaction with the breasts and self-esteem on BII risk are evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Floor van Leeuwen, PhD, Principal Investigator — The Netherlands Cancer Institute; Marie-Jeanne Vrancken Peeters, PhD, Principal Investigator — The Netherlands Cancer Institute; Eveline Bleiker, Principal Investigator — The Netherlands Cancer Institute
Locations (7):
- Netherlands (7):
  - Zuyderland Medical Center, Heerlen, Limburg
  - Maastricht University Medical Center, Maastricht, Limburg
  - Netherlands Cancer Institute Antoni van Leeuwenhoek, Amsterdam, North Holland
  - Velthuis Kliniek, Hilversum, North Holland
  - Ziekenhuisgroep Twente, Almelo, Overijssel
  - Medisch Spectrum Twente, Enschede, Overijssel
  - Erasmus MC University Medical Center, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Spoor J, de Jong D, van Leeuwen FE. [Silicone breast implants: the importance of nuanced reporting]. Ned Tijdschr Geneeskd. 2022 Mar 21;166:D6515. Dutch. PMID 35499539
- [Background] Spoor J, de Jong D, van Leeuwen FE. Silicone Particle Migration: A Misleading Report. Aesthet Surg J. 2022 Mar 15;42(4):NP261-NP262. doi: 10.1093/asj/sjab377. No abstract available. PMID 34695179
- [Derived] Spoor J, Mureau MAM, Tissier RLM, Hommes J, Rakhorst H, de Boer M, Oldenburg HSA, Heuts EM, Vissers YLJ, Dassen AE, Evers DJ, Koppert LB, Zaal LH, Linn SC, de Jong D, van der Hulst RRWJ, Vrancken Peeters MTFD, Bleiker EMA, van Leeuwen FE. Breast implant illness after reconstruction with silicone breast implants. J Natl Cancer Inst. 2025 Aug 1;117(8):1717-1728. doi: 10.1093/jnci/djaf136. PMID 40605595
- [Derived] Spoor J, Mureau MAM, Hommes J, Rakhorst H, Dassen AE, Oldenburg HSA, Vissers YLJ, Heuts EM, Koppert LB, Zaal LH, van der Hulst RRWJ, Vrancken Peeters MTFD, Bleiker EMA, van Leeuwen FE; AREOLA Collaboration. The Areola study: design and rationale of a cohort study on long-term health outcomes in women with implant-based breast reconstructions. Ann Epidemiol. 2023 Jun;82:16-25. doi: 10.1016/j.annepidem.2023.04.001. Epub 2023 Apr 6. PMID 37028614
- See also: Website RIVM: Onderzoeksprogramma vrouwen met een siliconen borstimplantaat — https://www.rivm.nl/medische-hulpmiddelen/siliconen-borstimplantaten/onderzoeksprogramma-gezondheidsklachten